CLINICAL TRIAL: NCT04374396
Title: The Effect of Erector Spinea Plane Block on the Postoperative Analgesia in Pediatric Hip Surgery: Randomized Controlled Study
Brief Title: Erector Spinea Plane Block in Pediatric Hip Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sameh Abdelkhalik Ahmed Ismaiel, Assistant Professor of Anesthesia - Tanta Faculty of Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 33779/4/20
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Last update posted 2021-02-05 (Actual); Status verified 2021-02

CONDITIONS: Postoperative Pain; Opioid Use
Keywords: Erecto spinae plane; Hip surgery; Children; Pain; Morphine consumption
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Intervention Model Description: Parallel Assignment Prospective study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Sham ESP block will be administrated in the control group Measurements will be obtained by anesthetist not participating in the study and blinded to its group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Sham Comparator): patients in this group will receive sham ipsilateral ultrasound-guided single shot erector spinae block at L2 after induction of anaesthesia and before the start of surgery without injection of local anesthetics
  Interventions: Radiation: Sham ultrasound-guided single shot erector spinae plane block (ESP B)
- Group 2 (Experimental): patients in this group will receive real ipsilateral ultrasound-guided single shot erector spinae block at L2 after induction of anaesthesia and before the start of surgery with injection of 0.3 ml/kg of 0.25% of plain bupivacaine.
  Interventions: Procedure: Real ultrasound-guided single shot erector spinae plane block (ESP B)

INTERVENTIONS:
Procedure: Real ultrasound-guided single shot erector spinae plane block (ESP B) — ESP block will be performed with the patient lying in the lateral position and the surgical side at the top. After skin disinfection, sterile draping will be placed, and ultrasound probe will be sheathed. The level of the block will be at the transverse process of L2, using a 9-12 MHz linear probe and placed in a parasagittal plane 1 cm from the posterior midline. The deep plane to the erector spinae muscle (ESM) will be identified and a 22 Gauge 50 mm insulated needle will be inserted craniocaudally in plane between the transverse process and the fascia of the ESM.
  After negative aspiration, 0.3 mL/kg- of bupivacaine 0.25% will be injected confirming correct position by visualizing the solution lifting the ESM off the transverse process .Spread of LA between the L1 and L4 transverse processes will be thereafter visually tracked with the transducer. In the control group, no local anesthetics will be injected.
  Arms: Group 2
Radiation: Sham ultrasound-guided single shot erector spinae plane block (ESP B) — EESP block will be performed with the patient lying in the lateral position and the surgical side at the top. After skin disinfection, sterile draping will be placed, and ultrasound probe will be sheathed. The level of the block will be at the transverse process of L2, using a 9-12 MHz linear probe and placed in a parasagittal plane 1 cm from the posterior midline. The deep plane to the erector spinae muscle (ESM) will be identified and a 22 Gauge 50 mm insulated needle will be inserted craniocaudally in plane between the transverse process and the fascia of the ESM.
  No local anesthetics will be injected
  Arms: Group 1

SUMMARY:
This prospective randomized controlled double-blind study will be carried out to evaluate the effect of ultrasound-guided erector spinae plane block on the postoperative analgesia in children after hip surgeries, the total morphine consumption in the first postoperative day will be the primary outcome and the time to first request for rescue analgesia and postoperative pain score will be the secondary outcome.

The study will be carried out on pediatric patients undergoing hip surgery where they will receive real or sham ultrasound guided erector spinae plane block before the onset of the surgery.

DETAILED DESCRIPTION:
This prospective randomized controlled double-blind study will be carried out to evaluate the effect of ultrasound-guided erector spinae plane block on the postoperative analgesia in children after hip surgeries.

Primary outcome: Total morphine consumption in the first postoperative day. Secondary outcome: The time to first request for rescue analgesia and postoperative pain score.

This clinical trial will be carried out in Tanta University Hospitals for a period of 6 month that may be extended on pediatric patients scheduled for surgical treatment of hip disorder under general anesthesia.

A written informed consent will be obtained from the parents of all patients. Randomization will be performed by an independent data manager assigned the patients to groups based on a computer-generated randomization program introduced in closed opaque envelope.

Group 1 (20 patients): patients in this group will receive sham ipsilateral ultrasound-guided single shot erector spinae block at the level of second lumbar vertebra after induction of anesthesia and before the start of surgery without injection of local anesthetics.

Group 2 (20 patients): patients in this group will receive real ipsilateral ultrasound-guided single shot erector spinae block att the level of second lumbar vertebra after induction of anesthesia and before the start of surgery with injection of 0.3 ml/kg of 0.25% of plain bupivacaine.

Anesthetic technique All the patients will be adequately assessed preoperatively in the anesthesia clinic through history taking, general and local examination, and requesting investigation. Adequate explanation of the procedure, benefit, and potential hazards will be done to the parents with final reassurance of them. All children will receive sedation in the form of oral midazolam 0.5 mg/kg 15 minutes before admission to the operating room.

Upon admission to the operating room, intravascular access will be obtained with starting i.v infusion of Dextrose 5% in normal saline (7 ml/kg). Then, the patients will be attached to a monitor of pulse oximetry, non-invasive blood pressure, end-tidal carbon dioxide, temperature, and 5 leads electrocardiogram. Induction of anesthesia will be carried out using sevoflurane 6% in oxygen: air (4:1) till the child loss the consciousness, then, fentanyl 0.5 ug/kg will be given intravenously and atracurium 0.5 mg/kg will be given intravenously to facilitate endotracheal intubation. A suitable sized endotracheal tube will be introduced and secured with connection of the patients to a mechanical ventilator (pressure-controlled mode) which parameters will be adjusted to maintain end-tidal carbon dioxide 36-40 mmHg.

Anesthesia will be maintained by sevoflurane (1 MAC) with incremental doses of atracurium. Also, incremental doses of fentanyl 0.5 ug/kg will be given i.v in case of increase bispectral index (BIS) more than 60 or by increase in the heart rate or the mean arterial pressure by more than 20% of the baseline values.

ELIGIBILITY:
Inclusion Criteria:

* Children aged between 1-5 years old, of both sexes, American Society of Anesthesiologists (ASA) physical status class I-II and scheduled for surgical treatment of hip disorder under general anesthesia will be included in this study

Exclusion Criteria:

1. Parental refusal.
2. Preexisting spinal deformity or profound mental retardation.
3. Obese Children
4. Known or suspected allergy to local anesthetics.
5. Known or suspected coagulopathy
6. Major cardiac, renal, or hepatic disorders.
7. Children undergoing combined or bilateral surgeries.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-02-01 (Actual); Study Completion 2021-02-02 (Actual)

PRIMARY OUTCOMES:
Total morphine consumption in the first postoperative day | The first 24 hours after surgery
  Calculation of the total dose of morphine consumed in the first day after surgery

SECONDARY OUTCOMES:
The time to first request for rescue analgesia | The first 24 hours after surgery
  The time interval from the end of the surgery till the first dose of morphine administrated
Postoperative pain score | every 2 hours in the first 8 hours then every 4 hours till 24 hours
  The postoperative pain score (CHEOPS pain score)

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Ismaiel, M.D, Study Director — Lecturer of Anesthesia and Intensive Care, Tanta University; Mohamed Abdullah, M.D, Study Director — Assistant Professor of Anesthesia and Intensive Care, Tanta University
Locations (1):
- Faculty of Medicine, Tanta, Algharbia, Egypt

IPD SHARING:
Plan to Share IPD: No
Once the study had been successfully completed, the data will be shared for other researchers.